CLINICAL TRIAL: NCT02597387
Title: A Single-arm, Open, Multi-center Phase II Clinical Trial of Mitoxantrone HCL Liposome Injection in Subjects With Relapsed Diffuse Large B-cell Lymphoma and and Peripheral T/NK Lymphomas
Brief Title: Clinical Trial of Mitoxantrone HCL Liposome Injection in Patients With Relapsed DLBCL and PT/NKCLs
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-HE153/PRO/Ⅱ
Record Dates: First submitted 2015-11-03; First posted 2015-11-05 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-05

CONDITIONS: Relapsed DLBCL and PT/NKCLs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mitoxantrone HCL Liposome Injection (Experimental): Each treatment cycle lasts for 28 days with 20mg/m2
  Interventions: Drug: Mitoxantrone HCL Liposome Injection

INTERVENTIONS:
Drug: Mitoxantrone HCL Liposome Injection

SUMMARY:
To study efficacy and safety of Mitoxantrone HCL Liposome Injection in patients with diffuse large B-cell lymphoma and lymphoma peripheral T cell.

DETAILED DESCRIPTION:
A Single-arm, Open, Multi-center Phase II Clinical Trial of Mitoxantrone HCL Liposome Injection in Subjects With Relapsed Diffuse Large B-cell Lymphoma and and Peripheral T/NK Lymphomas with dose of 20 mg/m2.

ELIGIBILITY:
Inclusion Criteria:

* The subjects are voluntary and sign the informed consent form;
* ECOG score 0 to 2;
* The expected survival time ≥3 months;
* Diffuse large B-cell and peripheral T/NK cell non-Hodgkin's lymphomas confirmed with histopathology, and the peripheral T/NK cell lymphomas that are only limited to the following types: peripheral T-cell lymphoma (not otherwise specified), angioimmunobl;
* Failure or relapse after at least once of systemic treatment, and patients who can not receive autologous peripheral blood stem cell transplantation
* The major diameter of a single measurable lesion ≥1.5 cm in at least one measurable lesion;
* An interval of at least four weeks after the target tumor was treated with chemotherapy, radiotherapy, biological therapy, stem cell transplantation or other study drugs;
* Subjects at childbearing age agree to take effective contraceptive measures during the study; blood pregnancy test result is negative (except infertility due to menopause or operation);
* Laboratory tests (blood routine, liver and kidney function) meet the following requirements:

  * ANC≥ 1.5×109/L, for those with bone marrow involvement, ANC ≥ 1.0×109/L;
  * PLT ≥ 75×109/L, for those with bone marrow involvement, PLT ≥ 50 × 109/L;
  * Hb ≥ 9 g/dL; d) Cr) ≤ 1.5x ULN ;
  * TBIL ≤ 1.5x ULN;
  * AST or ALT ≤2.5 x ULN (for patients with liver metastases, ≤ 5 x ULN ).

Exclusion Criteria:

* Pregnant or lactating women;
* An allergic history to anthracyclines or liposome drugs;
* Disease progression or recurrence after anthracycline treatment within six months before the enrollment;"
* Patients who once used mitoxantrone injection;
* Patients who have used doxorubicin (or pirarubicin) with the total cumulative dose> 360mg/m2, or epirubicin with the total cumulative dose > 600mg/m2;
* Left ventricular ejection fraction is < 50% or < the lower limit of normal; clinically significant QT interval prolongation (>450ms in male, >470ms in female); a past history of cardiac disease caused by anthracyclines; a history of severe heart disease;
* Concomitant treatment as other anticancer drugs are needed;
* Lymphoma involving the central nervous system;
* Clinically active infection that can significantly affect the clinical trial;
* Within 6 weeks after organ transplantation or major organ surgery;
* Those who are inappropriate to be enrolled as evaluated by the researchers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-08; Primary Completion 2018-09 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR; complete response + partial response [CR + PR]) | Up to 6 months

SECONDARY OUTCOMES:
Duration of Response (DOR) | Time from the date at which the patient's objective status is first noted to be a CR or PR to the earliest date progression is documented (assessed up to approximately 24 months)
Time to Response (TTR) | Time from the date of registration to the date at which the patient's objective status is first noted to be a CR or PR (assessed up to approximately 24 months)
Progression-free survival (PFS) | Up to a total of 24 months after first dose or until disease progression, withdrawal from study, or death

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhu, Ph.D, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, China